CLINICAL TRIAL: NCT00058890
Title: Study of Gabapentin for the Pruritus of Cholestasis
Brief Title: Gabapentin to Treat Itch in Patients With Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R03 --9618 (completed 2005); R03DK055618 (NIH)
Record Dates: First submitted 2003-04-14; First posted 2003-04-16 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Liver Disease; Cholestasis; Cirrhosis; Pruritus; Itching
Keywords: itching; pruritus; cholestasis; liver disease; hepatitis; cirrhosis
MeSH Terms: conditions — Liver Diseases; Cholestasis; Fibrosis; Pruritus; Hepatitis | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Experimental)
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Under code, the study drug was started at 100 mg by mouth 3 times a day for 3 days, to be increased, if necessary and in the absence of side effects, by 300 mg every 3 days to a maximum of 2,400 mg daily in divided doses.
  Arms: Gabapentin
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this study, the effect of the medication gabapentin to treat itching secondary to liver disease is being studied.

There are some funds to cover travel expenses for patients who are not from New York (NY).

Gabapentin is approved to treat seizures in human beings. In this study, patients with liver disease who meet inclusion criteria are admitted to the research hospital of the New York Presbyterian Hospital to record scratching behavior by the use of a machine designed for that purpose. Blood work will be obtained. After completion of recording, patients are assigned by chance to receive active medication or placebo (a capsule that does not contain active medication). The patients will come to the outpatient office of the research hospital 2 weeks into the study for an interview and blood work. After 4 weeks, patients are readmitted to the hospital to record scratching behavior. After data are collected, the code is broken, if patient had been on inactive drug, active drug will be supplied as per protocol for 4 weeks. Blood work will be obtained. If patient had been randomized to active medication, the study will provide one week supply of drug. After that, the referring physician, with whom the study was previously discussed, could prescribe the medication as it is available.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled study of gabapentin for the pruritus of cholestasis. Duration: 4 weeks. Some travel funds available for patients from out of the NY area for all the visits. Hospitalization at baseline and after 4 weeks of treatment. One outpatient department visit at week 2.

All patients have to be referred by their physician, who will receive a summary of the results at the end of the patient's study participation.

If patients are randomized to active drug and respond to it with decrease in pruritus, a one week supply of medication is given. The referring physician could prescribe the drug for long term use. If the patient is randomized to placebo they can be treated with active medication provided by the study for 4 weeks, at end of which, the drug could be prescribed by referring physician if the patient responds to the drug with decrease in the pruritus.

ELIGIBILITY:
Inclusion criteria include:

* Patients from ages 18 to 80 with chronic pruritus secondary to liver disease

Patients must have:

* a normal chest X- ray during the previous year
* normal thyroid function tests (treated thyroid dysfunction is acceptable)
* controlled diabetes, if diabetes mellitus is present
* negative fecal occult blood within the previous year

Exclusion criteria include:

* history of hepatic encephalopathy
* decompensated liver disease as suggested by ascites and history of variceal bleeding
* malignancy
* inability to practice contraception
* pregnancy
* creatinine > 1.7 mg/dl
* hemoglobin < 10mg/dl
* S/P liver transplantation
* HIV infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-11 (Actual); Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Change in scratching activity monitoring system | 4 weeks
  A scratching activity monitoring system specifically designed to record scratching behavior independent of gross body movement

SECONDARY OUTCOMES:
Change in visual analogue scale for pruritus | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nora V Bergasa, M.D., Principal Investigator — New York Presbyterian Hospital Columbia University College of Physicians and Surgeons
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States

REFERENCES:
- [Result] Bergasa NV, McGee M, Ginsburg IH, Engler D. Gabapentin in patients with the pruritus of cholestasis: a double-blind, randomized, placebo-controlled trial. Hepatology. 2006 Nov;44(5):1317-23. doi: 10.1002/hep.21370. PMID 17058231